CLINICAL TRIAL: NCT05730790
Title: Immersive Virtual Reality for Dual-task Training in Older Adults With Mild Cognitive Impairment: A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tan Tock Seng Hospital (Other)
Collaborators: Nanyang Polytechnic (Other); National Neuroscience Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020/00262
Record Dates: First submitted 2023-02-02; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Block randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive-motor dual task training (DTT) (Experimental): Participants attended 14 sessions (40 minutes each) of dual task cognitive-motor training, 2 times per week for 7 weeks. Each cognitive-motor training session comprised of performing a dual task activity - gameplay using a virtual reality (VR) system while walking on a treadmill, of progressive difficulty pitched to the participant's performance.
  Interventions: Other: Cognitive-motor dual task training (DTT)
- Cognitive single task training (CSTT) (Active Comparator): Participants attended 14 sessions (32 minutes each) of single task cognitive training, 2 times per week for 7 weeks. Each cognitive training session comprised of game play using a virtual reality (VR) system, of progressive difficulty pitched to the participant's performance
  Interventions: Other: Cognitive single task training (CSTT)
- Motor single task training (MSTT) (Active Comparator): Participants attended 14 sessions (40 minutes each) of single task motor training over a period of 7 weeks. Each motor training session comprised of walking on a treadmill, of progressive difficulty pitched to the participant's performance
  Interventions: Other: Motor single task training (MSTT)

INTERVENTIONS:
Other: Cognitive-motor dual task training (DTT) — For session 1 to 3, the training comprises of 4 cycles of the following: 2 min dual tasking, 2 min rest, 2 min dual tasking, 2 min rest. For session 4 to 6, the training comprises of 4 cycles of the following: 2.5 min dual tasking, 1.5 min rest, 2.5 min dual tasking, 1.5 min rest. For session 7 to 14, the training comprises of 4 cycles of the following: 3 min dual tasking, 1 min rest, 3 min dual tasking, 1 min rest. The treadmill speed is maintained at 40%, 50% and 60% of participant's original gait speed at session 1 to 3, 4 to 6, and 7 to 14 respectively.
  There are 10 levels in the VR game. Participant will start at level 1 of VR game at session 1 and can progress to the next level at the subsequent session if game percentage > 80%.
  Arms: Cognitive-motor dual task training (DTT)
Other: Cognitive single task training (CSTT) — For session 1 to 3, the training comprises of 4 cycles of the following: 2 min VR gaming, 2 min rest, 2 min VR gaming and 2 min rest. For session 4 to 6, the training comprises of 4 cycles of the following: 2.5 min VR gaming, 1.5 min rest, 2.5 min VR gaming and 1.5 min rest. For session 7 to 14, the training comprises of 4 cycles of the following: 3 min VR gaming, 1 min rest, 3 min VR gaming and 1 min rest.
  There are 10 levels in the VR game. Participant will start at level 1 of VR game at session 1 and can progress to the next level at the subsequent session if game percentage > 80%.
  Arms: Cognitive single task training (CSTT)
Other: Motor single task training (MSTT) — For session 1 to 3, the training comprises of 4 cycles of the following: 8 min treadmill walking at 40% of participant's original gait speed followed by 2 min rest. For session 4 to 6, the training comprises of 4 cycles of the following: 8 min treadmill walking at 50% of participant's original gait speed followed by 2 min rest. For session 7 to 14, the training comprises of 4 cycles of the following: 8 min treadmill walking at 60% of the participant's original gait speed followed by 2 min rest.
  Arms: Motor single task training (MSTT)

SUMMARY:
Mild cognitive impairment (MCI) is a pre-dementia state marked by a higher risk of conversion to dementia. Presently, strategies to delay the progression of MCI to dementia, such as routine exercise and cognitive activities, are limited and only moderately efficacious. Cognitive-motor dual task training, enhanced in a virtual reality environment, is a novel intervention for individuals with MCI.

DETAILED DESCRIPTION:
A randomized controlled trial will be conducted. 54 patients with MCI will be recruited from an outpatient clinic. The participants will be randomly allocated to one of the three study arms. All three groups will participate in 2 training sessions per week for 7 weeks. Each session lasts 32 to 40 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 - 80 years of age
* Diagnosis of mild cognitive impairment (MCI)
* Able to walk independently without assistance, whether from a person or a walking aid

Exclusion Criteria:

* Diagnosed dementia (at the point of recruitment)
* Presence of end stage lung, cardiac, liver and/or renal disease
* Unstable acute medical conditions that prevent one from exercising on a treadmill
* Presence of active arthritis, with symptoms affecting function
* Cerebrovascular and/or cardiac events in the last 6 months
* Parkinson's disease
* History of hip fracture within the last 6 months
* History of epilepsy with seizures in the last 2 years
* Poor vision, not correctable by glasses
* Hearing difficulty (if unable to hear well at normal conversational volume)
* Acute backache with pain affecting ambulation
* Acute lower limb pain with pain affecting ambulation
* Cervical spondylosis with myelopathy or cervical spine issues
* Chronic vertigo
* Vestibular problems, causing issues with balance

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in dual-task gait cost measured using Optogait | Baseline, post-intervention after session 14 (week 7), 6 month
  Gait parameters collected include step length, single support time, double support time, step time, stride length, speed and cadence. Gait parameters are collected under both single and dual-task (serial seven subtraction and animal naming) conditions.
  Dual-task cost calculated as 100*(single task parameter - dual-task parameter)/single task parameter
Change in dual-task cognitive cost measured using corrected response rate of cognitive tasks | Baseline, post-intervention after session 14 (week 7), 6 month
  Cognitive tasks include 30 seconds serial seven subtraction and animal naming, under both single and dual-task conditions (while walking)

SECONDARY OUTCOMES:
Change in number of falls measured using a falls diary | Baseline, 6 month
  Number of falls in the past 12 months
Change in balance parameters and falls risk measured using Berg Balance Scale (BBS) | Baseline, post-intervention after session 14 (week 7), 6 month
  BBS is a 14-item tool which objectively assesses static balance and falls risk.
Change in falls risk measured using Timed Up and Go test (TUG) | Baseline, post-intervention after session 14 (week 7), 6 month
  TUG is a evaluative tool which assesses functional mobility and falls risk
Change in falls concerns scored using the Falls Efficacy Scale International (FES-I) | Baseline, post-intervention after session 14 (week 7), 6 month
  FES-I is a 16-item questionnaire used to measure the level of concern about falling during social and physical activities.
Change in executive function measured using Chinese Frontal Assessment Battery | Baseline, 6 month
  CFAB is brief tool used to assess frontal dysfunction via a series of neuropsychological tasks. A higher score indicates better performance with a total maximum of 18.
Change in executive function scored using the Stroop color-word test - Victoria version (VST) | Baseline, 6 month
  VST assess executive functioning using three conditions that consist in naming color of dots, of neutral words, and of color words printed in incongruent colors.
Change in sustained and divided attention assessed using Color Trails Test 1 and 2 | Baseline, 6 month
  Color Trails Test is the language free version of Trails Making Test, developed for cross-cultural assessment of sustained and divided attention in adults

CONTACTS AND LOCATIONS:
Overall Officials: Kwee Yong Joyce Yap, M.B.B.S., Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perez-Marcos D, Bieler-Aeschlimann M, Serino A. Virtual Reality as a Vehicle to Empower Motor-Cognitive Neurorehabilitation. Front Psychol. 2018 Nov 2;9:2120. doi: 10.3389/fpsyg.2018.02120. eCollection 2018. PMID 30450069
- [Background] Schwenk M, Zieschang T, Oster P, Hauer K. Dual-task performances can be improved in patients with dementia: a randomized controlled trial. Neurology. 2010 Jun 15;74(24):1961-8. doi: 10.1212/WNL.0b013e3181e39696. Epub 2010 May 5. PMID 20445152
- [Background] Muir SW, Speechley M, Wells J, Borrie M, Gopaul K, Montero-Odasso M. Gait assessment in mild cognitive impairment and Alzheimer's disease: the effect of dual-task challenges across the cognitive spectrum. Gait Posture. 2012 Jan;35(1):96-100. doi: 10.1016/j.gaitpost.2011.08.014. Epub 2011 Sep 22. PMID 21940172
- [Background] Fritz NE, Cheek FM, Nichols-Larsen DS. Motor-Cognitive Dual-Task Training in Persons With Neurologic Disorders: A Systematic Review. J Neurol Phys Ther. 2015 Jul;39(3):142-53. doi: 10.1097/NPT.0000000000000090. PMID 26079569
- [Background] Montero-Odasso MM, Sarquis-Adamson Y, Speechley M, Borrie MJ, Hachinski VC, Wells J, Riccio PM, Schapira M, Sejdic E, Camicioli RM, Bartha R, McIlroy WE, Muir-Hunter S. Association of Dual-Task Gait With Incident Dementia in Mild Cognitive Impairment: Results From the Gait and Brain Study. JAMA Neurol. 2017 Jul 1;74(7):857-865. doi: 10.1001/jamaneurol.2017.0643. PMID 28505243
- [Background] Delbroek T, Vermeylen W, Spildooren J. The effect of cognitive-motor dual task training with the biorescue force platform on cognition, balance and dual task performance in institutionalized older adults: a randomized controlled trial. J Phys Ther Sci. 2017 Jul;29(7):1137-1143. doi: 10.1589/jpts.29.1137. Epub 2017 Jul 15. PMID 28744033
- [Background] Camicioli R, Howieson D, Lehman S, Kaye J. Talking while walking: the effect of a dual task in aging and Alzheimer's disease. Neurology. 1997 Apr;48(4):955-8. doi: 10.1212/wnl.48.4.955. PMID 9109884
- [Background] Mirelman A, Rochester L, Reelick M, Nieuwhof F, Pelosin E, Abbruzzese G, Dockx K, Nieuwboer A, Hausdorff JM. V-TIME: a treadmill training program augmented by virtual reality to decrease fall risk in older adults: study design of a randomized controlled trial. BMC Neurol. 2013 Feb 6;13:15. doi: 10.1186/1471-2377-13-15. PMID 23388087
- [Background] Verghese J, Wang C, Lipton RB, Holtzer R. Motoric cognitive risk syndrome and the risk of dementia. J Gerontol A Biol Sci Med Sci. 2013 Apr;68(4):412-8. doi: 10.1093/gerona/gls191. Epub 2012 Sep 17. PMID 22987797
- [Background] Abdin E, Subramaniam M, Achilla E, Chong SA, Vaingankar JA, Picco L, Sambasivam R, Pang S, Chua BY, Ng LL, Chua HC, Heng D, Prince M, McCrone P. The Societal Cost of Dementia in Singapore: Results from the WiSE Study. J Alzheimers Dis. 2016;51(2):439-49. doi: 10.3233/JAD-150930. PMID 26890766